CLINICAL TRIAL: NCT01902264
Title: Prospective, Open-label, Single-center Clinical Study to Investigate the Red Blood Cell and Plasma Folate Concentrations During a 24-week Treatment Period With the Combination of Drospirenone 3 mg Plus Ethinyl Estradiol 0.02 mg Plus Levomefolate Calcium 0.451 mg in Mexican Women Seeking Contraception
Brief Title: Study of Treatment With the Combination of Drospirenone Plus Ethinyl Estradiol Plus Levomefolate Calcium in Mexican Women Seeking Contraception
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16484
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Contraception
Keywords: Levomefolate calcium; Contraceptives, oral, combined; Neural tube defects
MeSH Terms: conditions — Neural Tube Defects | interventions — beyaz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EE20/DRSP/L-5-MTHF (Experimental)
  Interventions: Drug: EE20/DRSP/L-5-MTHF (Beyaz, BAY98-7071)

INTERVENTIONS:
Drug: EE20/DRSP/L-5-MTHF (Beyaz, BAY98-7071) — One tablet DRSP 3 mg/EE 0.02 mg/ Levomefolate calcium 0.451 mg daily for 24 days, followed by one hormone-free tablet L-5-MTHF 0.451 mg daily for 4 days over 24 weeks

SUMMARY:
The objective of this study is to compare the red blood cell (RBC) and plasma concentrations of folate in subjects treated with drospirenone (DRSP)/ethinyl estradiol (EE) plus levomefolate calcium (L-5-MTHF) at 24 weeks with respect to basal determination.

Increased intake of folic acid (synthetic form of the naturally occurring B-vitamin) before and in the first few weeks of pregnancy has been shown to reduce certain types of birth defects. This is important for women who may become pregnant following discontinuation of oral contraception. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Mexican female subjects requesting contraception
* Age >/=18 to </=45 years (inclusive); smokers must not be older than 30 years at the time of informed consent
* Normal or clinically insignificant cervical smear not requiring further follow-up; a cervical smear has to be taken at the screening visit, or a normal result has to be documented within the previous 6 months. Human papilloma virus (HPV) testing in subjects with atypical squamous cells of undetermined significance (ASCUS) can be used as an adjunctive test. Subjects with ASCUS can be included if they are negative for high-risk HPV strains.

Exclusion Criteria:

* Pregnancy or lactation (less than 6 months since delivery, abortion, or lactation before start of treatment)
* Body mass index (BMI) >30 kg/m2
* Hypersensitivity to any ingredient in the study drug
* Any diseases or conditions that can compromise the function of body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study medication
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Any disease or condition that may worsen under hormonal treatment according to the assessment and opinion of the investigator.
* Undiagnosed abnormal genital bleeding
* Abuse of alcohol, drugs or medicine (eg, laxatives)
* Any medication that could result in excessive accumulation, impaired metabolism, or altered excretion of the study drug

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in RBC folate concentration from baseline to Week 24 | Baseline and Week 24
Change in plasma folate concentration from baseline to Week 24 | Baseline and Week 24

SECONDARY OUTCOMES:
RBC folate concentration | Different time points up to 32 weeks
Plasma folate concentration | Different time points up to 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mexico City, Mexico City, Mexico